CLINICAL TRIAL: NCT05892757
Title: A Phase 1 Lactation Study in Healthy Adult Lactating Female Subjects One to Six Months Post-Partum to Evaluate the Pharmacokinetics and Safety of Ubrogepant and Atogepant
Brief Title: Study to Assess Adverse Events and Compare How Oral Ubrogepant and Oral Atogepant Moves Through the Body of Healthy Female Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M22-394
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Atogepant; Ubrogepant
MeSH Terms: interventions — atogepant; ubrogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atogepant (Experimental): Participants will receive single dose of atogepant on Day 1.
  Interventions: Drug: Atogepant
- Ubrogepant (Active Comparator): Participants will receive single dose of ubrogepant on Day 1.
  Interventions: Drug: Ubrogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA
  Arms: Atogepant
Drug: Ubrogepant — Oral Tablet
  Other Names: UBRELVY
  Arms: Ubrogepant

SUMMARY:
This study will assess adverse events and compare how ubrogepant and atogepant tablets move through the body of healthy adult lactating female participants.

Ubrogepant and atogepant are approved drugs for treatment of migraine in adults. Participants will be assigned to one of the 2 treatment arms to receive atogepant or ubrogepant. Approximately 24 healthy adult lactating female participants will be enrolled at 3 sites in the United States

Participants will receive oral tablets of ubrogepant or atogepant on Day 1 and will be followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, lactating, female volunteers who delivered one or more normal-term infants and established lactation from 1 - 6 months post-partum at the time of enrollment.
* Had a normal pregnancy (gestation of 37-42 weeks) with no clinically significant complications.
* Willing to permit the use of pasteurized donor milk, infant formula, or previously pumped/stored human milk to feed the infant.
* Agree to the use of provided breast pumps for the pumping of breast milk during the milk collection regimen of the study.

Exclusion Criteria:

- Prior exposure to ubrogepant or atogepant within the past 30 days.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to Day 30
  An adverse event is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Plasma Concentration (Cmax) of Atogepant | Up to Day 2
  Cmax of Atogepant
Maximum Observed Plasma Concentration (Cmax)of Ubrogepant | Up to Day 2
  Cmax of Ubrogepant
Time to Cmax (Tmax) of Atogepant | Up to Day 2
  Tmax of Atogepant
Time to Cmax (Tmax) of Ubrogepant | Up to Day 2
  Tmax of Ubrogepant
Apparent Terminal Phase Elimination Rate Constant (β) of Atogepant | Up to Day 2
  Apparent terminal phase elimination rate constant of Atogepant
Apparent Terminal Phase Elimination Rate Constant (β) of Ubrogepant | Up to Day 2
  Apparent terminal phase elimination rate constant of Ubrogepant
Terminal Phase Elimination Half-life (t1/2) of Atogepant | Up to Day 2
  T1/2 of Atogepant
Terminal Phase Elimination Half-life (t1/2) of Ubrogepant | Up to Day 2
  T1/2 of Ubrogepant
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUCt) of Atogepant | Up to Day 2
  AUCt of Atogepant
AUCt of Ubrogepant | Up to Day 2
  AUCt of Ubrogepant
AUC From Time 0 to the Time Infinity (AUCinf) of Atogepant | Up to Day 2
  AUCinf of Atogepant
AUCinf of Ubrogepant | Up to Day 2
  AUCinf of Ubrogepant
Maximum Observed Breast Milk Concentration (CMAX) of Atogepant | Up to Day 2
  CMAX of Atogepant
Maximum Observed Breast Milk Concentration (CMAX) of Ubrogepant | Up to Day 2
  CMAX of Ubrogepant
Time to Maximum Observed Breast Milk Concentration (TMAX) of Atogepant | Up to Day 2
  TMAX of Atogepant
Time to Maximum Observed Breast Milk Concentration (TMAX) of Ubrogepant | Up to Day 2
  TMAX of Ubrogepant
Area Under the Milk Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUCLST) of Atogepant | Up to Day 2
  AUCLST of Atogepant
Area Under the Milk Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUCLST) of Ubrogepant | Up to Day 2
  AUCLST of Ubrogepant
Area Under the Milk Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCINF) of Atogepant | Up to Day 2
  AUCINF of Atogepant
Area Under the Milk Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCINF) of Ubrogepant | Up to Day 2
  AUCINF of Ubrogepant

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Bio-Kinetic Clinical Applications, LLC /ID# 255452, Springfield, Missouri
  - Icon /Id# 257524, San Antonio, Texas
  - Icon /Id# 257525, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boinpally RR, Smith JH, De Abreu Ferreira RL, Trugman JM. Pharmacokinetics of Atogepant in Healthy Lactating Female Participants: Results from a Phase 1 Lactation Study. Neurol Ther. 2025 Aug;14(4):1461-1473. doi: 10.1007/s40120-025-00772-4. Epub 2025 Jun 2. PMID 40455369
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-394